CLINICAL TRIAL: NCT07147907
Title: Respiratory Rate Validation Study
Status: Completed | Type: Observational
Sponsor: Perin Health Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: PR 2025-644
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Respiration Rate; Monitoring, Physiologic
Keywords: Respiratory rate validation; Breathing rate measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Chest Worn Respiratory Rate Monitor — The Perin Health Patch is a non-invasive, chest-worn wearable device designed to continuously monitor physiological signals, including respiratory rate and other health metrics. In this study, the device will be evaluated for its ability to accurately measure respiratory rate during controlled breathing exercises in healthy adult volunteers. The respiratory rate values recorded by the Perin Health Patch will be compared against respiratory rate measurements obtained via manually scored end tidal carbon dioxide (EtCO2) waveforms from a GE Datex-Ohmeda monitor, following Element Laboratory protocols aligned with clinical validation standards. The intervention in this study is limited to the application and use of the device for data collection during controlled respiratory rate conditions, where participants perform paced breathing exercises at various rates (5-50 breaths per minute) using a breathing app while positioned sitting or lying supine.

SUMMARY:
The goal of this clinical trial is to test how accurately a new chest-worn device called the Perin Health Patch measures breathing rate in adults aged 22 and older. The main question it aims to answer is:

How accurately does the Perin Health Patch measure breathing rate compared to a standard medical device that measures carbon dioxide in exhaled breath?

Participants will:

* Wear the Perin Health Patch on their chest during the study session
* Breathe through a mouthpiece or nose tube connected to a standard breathing monitor
* Follow guided breathing exercises at different speeds (from very slow to fast breathing) using a breathing app
* Sit and lie down in different positions during the measurements
* Complete the study in one visit lasting about 1-2 hours

The study will include both healthy adults and people with conditions like asthma, COPD, heart failure, diabetes, high blood pressure, or obesity to test how well the device works for different types of people. Researchers will compare the breathing rate numbers from the new chest patch to the standard medical device to see if the patch is accurate enough for medical use.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have the ability to understand and provide written informed consent.
* Participants or legally authorized representative must be able to read or write in English.
* Participant is adult, ages 22 years or older.
* Participant must be willing and able to comply with study procedures and duration.

Exclusion Criteria:

* Participant unwilling or unable to provide written informed consent.
* Participants evaluated by the Investigator and/or Clinical Staff and found to be medically unsuitable or have self-reported health conditions that are currently unstable as identified in Health Assessment Form and Health Screening.
* Compromised circulation, injury, or physical malformation of the fingers, toes, hands, ears or forehead/skull or other sensor ROI, which would limit the ability to test ROI.
* Tattoos in the optical path, which would limit the ability to test ROI. Certain malformations may still allow participants to participate if the condition is noted and would not affect the ROI.
* Participants with severe contact allergies to standard adhesives, latex, or other materials found in pulse oximeters, ECG electrodes, or other medical sensors (self-reported).
* Any other known health conditions may be evaluated and should be considered upon disclosure in health assessment form.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of a minimum of 35 adult participants and maximum of 80 adult participants, ages 22 years and older. The study population will be comprised of diversity in race, age, gender, BMI, skin tone, and health conditions. The health conditions will constitute certain proportions of healthy controls (to allow testing over the full range of breaths per minute) and disease comorbidities (to represent comorbidities such as COPD, CHF, Asthma, Diabetes, Hypertension, Diabetes and Obesity). An attempt will be made to enroll a variety of skin tones. The participants must understand the study and consent to participate by signing the Informed Consent Form. Participant enrollment and participation in this clinical study is based on meeting the inclusion criteria and none of the exclusion criteria, a satisfactory health screen, and the participant and data demographics needed for the study.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Accuracy of Perin Health Patch Respiratory Rate Measurements Compared to End Tidal CO₂ Reference | During a single in-lab session lasting approximately 1 hour per participant
  The primary outcome is the accuracy of respiratory rate (RR) values reported by the Perin Health Patch compared to respiratory rate measured by manually scored end tidal carbon dioxide (EtCO₂) waveforms from a GE Datex-Ohmeda monitor. Accuracy will be assessed using mean absolute error (MAE), accuracy root mean square (ARMS), bias (mean difference), and standard deviation. Measurements will be collected during multiple stable respiratory rate plateaus (approximately 5-50 breaths per minute) achieved through paced breathing exercises. Each comparison will be made during 60-second intervals at steady-state conditions, with the reference EtCO₂ waveform scored by blinded reviewers counting respiratory peaks per minute.

CONTACTS AND LOCATIONS:
Locations (1):
- Element Boulder, Louisville, Colorado, United States